CLINICAL TRIAL: NCT01485913
Title: A Randomized Trial of an Intensive Education Intervention Using a Network of Involved Diabetic Patients (Peer Educators) to Improve Glycemic Control of Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sante Diabete Mali (Other)
Collaborators: Bridges program, International Diabetes Federation (Unknown)
Responsible Party: Principal Investigator, Besancon Stephane, Director NGO Santé diabète, Sante Diabete Mali
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SDMBRIDGES01
Record Dates: First submitted 2011-07-20; First posted 2011-12-06 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Diabetes
Keywords: Education; Diabetes; Prevention complications; Prevention of complications of diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The methodologist who performed the randomisation was not directly involved in the recruitment of patients. Recruiting physicians were blinded to the allocation sequence.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Experimental): The group subjected to educations will follow the whole process of peer education described in Part 1 of this Protocol.
  The control group will perform these "classic" individual consultations but will not follow the whole process of peer education.
  The classical management in diabetes consultations consists of:
  * A counselling session
  * A measure of blood glucose
  * A measurement of blood pressure
  * A measure of weight and size
  * A complete clinical examination
  * A prescription or a renewal of treatment (diabetes pills, insulin, IEC, statins etc ...)
  Interventions: Other: intensive education intervention using a network of involved diabetic patients (peer educators)
- No Lifestyle counseling (No Intervention): The group subjected to educations will follow the whole process of peer education described in Part 1 of this Protocol.
  The control group will perform these "classic" individual consultations but will not follow the whole process of peer education.
  The classical management in diabetes consultations consists of:
  * A counselling session
  * A measure of blood glucose
  * A measurement of blood pressure
  * A measure of weight and size
  * A complete clinical examination
  * A prescription or a renewal of treatment (diabetes pills, insulin, IEC, statins etc ...)

INTERVENTIONS:
Other: intensive education intervention using a network of involved diabetic patients (peer educators) — the purpose of this methodology is to set up coordinated training and education activities targeting populations with diabetes based on a pragmatic approach (the learning nests methodology) of appropriation and construction of knowledge that takes into account the individual, social, economic, cultural context. This work is being implemented on the basis of group modules specifically designed in their running: are studied the concrete elements of knowledge to mobilize, patients' actions, the role of health the educator, indicators of progress and monitoring during sessions and on the long term. Each patient is gotten to consider the elements involved in his/her disease, and the actions that can be achieved taking into account the feasibility in his/her own context. The education monitoring is envisaged through a data compendium present in the individual booklets that are given to patients at the end of each education session.
  Arms: Lifestyle counseling

SUMMARY:
The project will test the implementation of a specific methodology for education of type 2 diabetic patients that will be set up using patients involved (peer educators) and 3 guides developed specifically for the therapeutic education of type 2 diabetic patients. This project will take place in 1 sites in mali : the capital Bamako. 75 diabetic patients will be subjected to intervention with this methodology and 75 other diabetic patients will be the control group. At various stages of the project, the investigators will analyze the impact on biological, anthropological constants, etc ... of the group undergoing the intervention compared to the control group.

DETAILED DESCRIPTION:
Title of project:

A randomized trial of an intensive education intervention using a network of involved diabetic patients (peer educators) to improve glycemic control of type 2 diabetic patients

Research question (s)/hypothesis:

Main objective of the research: compare the improvement of HbA1c 1 year after an intervention led by peer educators, versus a conventional care in health centre

Secondary objectives:

Study the evolution of bio clinical parameters: fasting glucose, weight, BMI, blood pressure, waist size

Method (s) :

This study will be conducted by a multidisciplinary team that brings together high level skills in research projects and in peer education projects. It will be conducted in one site in one country Mali.

This site was chosen because they meet a functional care, access to medicines and a dynamic association of diabetic patients. Peer educators and persons targeted by the project will be recruited through the local association of patients. This association will be a social support that provides on going prevention counseling, education and support services to people who have diabetes. It represents an important link between patients, educators and general medical services. The procedure will start by the training of peer educators who were identified and recruited to facilitate the sessions

Then, the 4 educational sessions: control of cardiovascular risk (blood pressure, waist circumference, smoking, cholesterol, glycaemia), control of Food (balance, fat, carbohydrates), physical activity management, insulin management, will be carried out and patients will be able to:

* Analyze knowledge that appears in various forms, including forms adapted to illiterate patients (colour codes, presence of photos)
* Act on knowledge: the patient observes, makes hypothesis, he experiments, compares, deduces, analyzes, makes relations.
* Work in interaction with other learners, which gives education a social dimension.
* Decide on the implementation of actions taking into account individual, cultural, social, economic context

For each situation, a day of training will be conducted by trained peer educators with theoretical contributions on the issue, practical scenarios, analyzes of the issues out of frame and put in "educational security ". These training days will be implemented with 8-10 patients (1Hour and an half) and the 4 sessions will take place over a period of two months starting from the inclusion of patients.

2 groups of 75 persons will be formed. One group will have specific education using methodology of learning nests. The other group will be a control group not subject to this specific education.

To evaluate, we propose a classical randomized controlled experimental (RCT) design, with randomization at the person-level. For outcome measures, we propose change in HbA1c, increase of social and emotional support and increase of linkage to clinical care. In addition to HbA1c, we propose measuring changes in systolic, diastolic blood pressure, and weight.

Public health significance (state how the project applies to your community and it potential impact(s))

It is very important to find an education methodology adapted to the African context. This line of diabetes management is essential to improve the management of African diabetic patients.

Sustainability plan:

If the evaluation of this methodology is conclusive, the Malian state will implement the methodology in the 22 diabetes units of the country.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed in the diabetes units of the project area and doing regular consultations
* Patients with type 2 diabetes or treated or not with insulin
* Poorly controlled diabetes with HbA1c ≥ 8%
* Patients who accepted to undergo the whole process of peer education
* Patients who agreed to perform all biological measures included in the protocol
* Patients aged from 30 to 80 years old

Exclusion Criteria:

* Diabetic patients not carrying out their monitoring in diabetes units of the intervention area
* Patients followed in the diabetes units of the intervention area but not realizing their consultations regularly
* Patients with type 1 diabetes
* Severe complications within the preceding 3 months: infection, coronary complications, severe renal failure
* Concomitant illnesses threatening the functional or vital prognosis

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2013-06-30 (Actual)

PRIMARY OUTCOMES:
Compare the intermediate evolution of the HbA1c (3, 6 and 12 months) | Change Hba1c from T0 to T12
  The main judgement criteria on which the analysis will be done to comply with the superiority of the contribution of a group educational approach by the peer will be the evolution of the HbA1c from the inclusion to 1 year.
  In practice the main measure is the measurement of glycated hemoglobin of patients expressed in %. We want to show that in the protocol by increasing the education of patients we're going to lower their HbA1c%

SECONDARY OUTCOMES:
Compare the evolution of the bio-clinical parameters at 3.6, and 12 months: weight, BMI, blood pressure, waist measurement | evolution at T = 0, 3 months, 6 months and 12 months of the systolic and diastolic blood pressure, weight, BMI and waist measurement.
  The secondary judgement criteria will be the evolution at T = 0, 3 months, 6 months and 12 months of the systolic and diastolic blood pressure, weight, BMI and waist measurement.
  In practice the secondaries measure is the measurement of blood pressure, size (m), weight (Kg) and weist mesurement (cm). We want to show that in the protocol by increasing the education of patients we're going to lower their blood pressure, BMI, weight and weist mesurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital National du Mali, Bamako, Mali

REFERENCES:
- [Derived] Debussche X, Besancon S, Balcou-Debussche M, Ferdynus C, Delisle H, Huiart L, Sidibe AT. Structured peer-led diabetes self-management and support in a low-income country: The ST2EP randomised controlled trial in Mali. PLoS One. 2018 Jan 22;13(1):e0191262. doi: 10.1371/journal.pone.0191262. eCollection 2018. PMID 29357380
- See also: Web site NGO Sante Diabète — http://www.santediabete.org